CLINICAL TRIAL: NCT00729586
Title: A Randomized Phase II Trial of Temsirolimus (NCI-Supplied Agent, NSC # 683864) or the Combination of Hormonal Therapy Plus Temsirolimus in Women With Advanced, Persistent, or Recurrent Endometrial Carcinoma
Brief Title: Temsirolimus With or Without Megestrol Acetate and Tamoxifen Citrate in Treating Patients With Advanced, Persistent, or Recurrent Endometrial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-01085; NCI-2009-01085 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); GOG-0248; CDR0000609740; GOG-0248 (Other: NRG Oncology); GOG-0248 (Other: CTEP); U10CA180868 (NIH); U10CA027469 (NIH)
Record Dates: First submitted 2008-08-06; First posted 2008-08-07 (Estimated); Results first posted 2018-08-27 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Endometrial Carcinoma; Recurrent Uterine Corpus Carcinoma; Stage IIIA Uterine Corpus Cancer; Stage IIIB Uterine Corpus Cancer; Stage IIIC1 Uterine Corpus Cancer; Stage IIIC2 Uterine Corpus Cancer; Stage IVA Uterine Corpus Cancer; Stage IVB Uterine Corpus Cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Megestrol Acetate; Tamoxifen; temsirolimus; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (temsirolimus) (Experimental): Patients receive temsirolimus IV over 30 minutes once weekly for 6 weeks. Courses repeat every 6 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Temsirolimus
- Arm II (temsirolimus, megestrol acetate, tamoxifen citrate) (Experimental): Patients receive temsirolimus as in Arm I and megestrol acetate PO BID for 3 weeks alternating with tamoxifen citrate PO BID for 3 weeks. Courses repeat every 6 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Megestrol Acetate; Drug: Tamoxifen Citrate; Drug: Temsirolimus

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Megestrol Acetate — Given PO
  Other Names: 17-Hydroxy-6-methylpregna-4,6-diene-3,20-dione acetate; 17.alpha.-Acetoxy-6-methylpregna-4,6-diene-3,20-dione; 6-Dehydro-6-methyl-17.alpha.-acetoxyprogesterone; 6-Methyl-6-dehydro-17.alpha.-acetoxyprogesterone; BDH 1298; BDH-1298; Maygace; Megace; Megestat; Megestil; Niagestin; Ovaban; Pallace; SC-10363
  Arms: Arm II (temsirolimus, megestrol acetate, tamoxifen citrate)
Drug: Tamoxifen Citrate — Given PO
  Other Names: Apo-Tamox; Clonoxifen; Dignotamoxi; Ebefen; Emblon; Estroxyn; Fentamox; Gen-Tamoxifen; Genox; ICI 46,474; ICI-46474; Jenoxifen; Kessar; Ledertam; Lesporene; Nolgen; Noltam; Nolvadex; Nolvadex-D; Nourytam; Novo-Tamoxifen; Novofen; Noxitem; Oestrifen; Oncotam; PMS-Tamoxifen; Soltamox; TAM; Tamax; Tamaxin; Tamifen; Tamizam; Tamofen; Tamoxasta; Tamoxifeni Citras; Zemide
  Arms: Arm II (temsirolimus, megestrol acetate, tamoxifen citrate)
Drug: Temsirolimus — Given IV
  Other Names: CCI-779; CCI-779 Rapamycin Analog; Cell Cycle Inhibitor 779; Rapamycin Analog; Rapamycin Analog CCI-779; Torisel

SUMMARY:
This randomized phase II trial studies how well temsirolimus with or without megestrol acetate and tamoxifen citrate works in treating patients with endometrial cancer that has spread to other places in the body and usually cannot be cured or controlled with treatment, has returned after a period of improvement, or is persistent. Temsirolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Estrogen can cause the growth of endometrial cancer cells. Hormone therapy using megestrol acetate and tamoxifen citrate may fight endometrial cancer by blocking the use of estrogen by the tumor cells. It is not yet known whether temsirolimus is more effective when given alone or together with megestrol acetate and tamoxifen citrate in treating endometrial cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the response rate of patients with advanced, persistent, or recurrent endometrial cancer when treated with each of the arms of the trial; the proposed arms are: Arm #1 temsirolimus intravenously (IV) weekly, Arm #2 megestrol (megestrol acetate)/tamoxifen (tamoxifen citrate) plus temsirolimus IV weekly.

II. Time to progression and number of patients remaining on study therapy at 24 weeks.

SECONDARY OBJECTIVE:

I. To describe the toxicities of each of the arms of the trial when used for patients with advanced/metastatic endometrial cancer.

TERTIARY OBJECTIVES:

I. Explore whether immunohistochemical expression of hormone receptors (estrogen receptor-alpha, estrogen receptor-beta, progesterone receptors-A, progesterone receptor-B and the alternative estrogen receptor, G protein-coupled estrogen receptor [GPR]-30) or components of the mammalian target of rapamycin (mTOR) signaling pathway (normal and mutant phosphatase and tensin homolog [PTEN], total and phosphorylated v-akt murine thymoma viral oncogene homolog 1 [Akt] as well as total and phosphorylated p70S6 kinase) are associated with treatment, outcome or clinical characteristics.

II. Explore whether single nucleotide polymorphisms (SNPs) in the FK506-binding protein 12-rapamycin-associated protein 1 (FRAP1) and regulatory associated protein of mTOR (RAPTOR) genes, mutations in phosphatidylinositol 4,5-bisphosphate 3-kinase catalytic subunit alpha (PIK3CA), PTEN and paxillin or copy number abnormalities in PTEN and paxillin are associated with treatment, outcome or clinical characteristics.

OUTLINE: Patients are randomized to 1 of 2 treatment arms. (Closed to accrual as of 11/22/2010)

ARM I: Patients receive temsirolimus IV over 30 minutes once weekly for 6 weeks. Courses repeat every 6 weeks in the absence of disease progression or unacceptable toxicity.

ARM II (Closed to accrual as of 12/21/2009): Patients receive temsirolimus as in Arm I and megestrol acetate orally (PO) twice daily (BID) for 3 weeks alternating with tamoxifen citrate PO BID for 3 weeks. Courses repeat every 6 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed advanced (International Federation of Gynecologists and Obstetricians [FIGO] stage III or IV), persistent, or recurrent endometrial carcinoma, which is not likely to be curable by surgery or radiotherapy; histologic documentation of the recurrence is not required
* All patients must have measurable disease; measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest dimension to be recorded); each lesion must be >= 20 mm when measured by conventional techniques, including palpation, plain x-ray, computed tomography (CT), and magnetic resonance imaging (MRI), or >= 10 mm when measured by spiral CT
* Patients must have at least one "target lesion" to be used to assess response, as defined by Response Evaluation Criteria In Solid Tumors (RECIST); tumors within a previously irradiated field will be designated as "non-target" lesions unless progression is documented
* Prior chemoradiotherapy for a pelvic recurrence is permitted; prior chemotherapy in the adjuvant setting for stage I, II, or III disease is permitted

  * Note: no prior chemotherapy in the setting of stage IV disease is permitted unless the patient was without evidence of disease at the completion of chemotherapy and had at least six months of progression-free survival since the completion of chemotherapy
  * Regardless of circumstances, no more than one prior chemotherapy regimen (including chemoradiotherapy) is permitted
* Patient must be able to take p.o. medications
* Performance status must be 0-2
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) =< 2.5 times institutional upper limit of normal v 3.0 (=< 5 times upper limit of normal [ULN] for subjects with liver metastases)
* Alkaline phosphatase =< 2.5 times institutional upper limit of normal v 3.0 (=< 5 times ULN for subjects with liver metastases)
* Creatinine =< 1.5 times normal institutional upper limit of normal
* Cholesterol =< 350 mg/dL (fasting)
* Triglycerides =< 400 mg/dL (fasting)
* Albumin >= 3.0 mg/dL
* At least 4 weeks must have elapsed since the patient underwent any major surgery (e.g., major: hysterectomy, resection of a lung nodule-minor: a Port-A-Cath placement)
* Patients who have met the pre-entry requirements
* Patients must have signed an approved informed consent including Health Insurance Portability and Accountability Act (HIPAA) authorization

Exclusion Criteria:

* Patients with Gynecologic Oncology Group (GOG) performance status of 3 or 4
* Patients cannot be receiving enzyme-inducing antiepileptic drugs (EIAEDs; e.g., phenytoin, carbamazepine, phenobarbital) nor any other cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) inducer such as rifampin or St. John's wort, as these may decrease temsirolimus levels; use of agents that potently inhibit CYP3A (and hence may raise temsirolimus levels), such as ketoconazole, is discouraged, but not specifically prohibited; the appropriateness of use of such agents is left to physician discretion

  * All concomitant medications must be recorded at baseline
* Patients on maintenance corticosteroids are ineligible with the exception of short term use (fewer than 5 days)
* Patients known to have congestive heart failure; patients with baseline requirement for oxygen; patients with serious concomitant illness that, in the opinion of the treating physician, will place patient at unreasonable risk from therapy on this protocol
* Patients with a history of unprovoked deep vein thrombosis (DVT) or pulmonary embolism (PE), unless patient is maintained on anticoagulation for the duration of the trial; while the exact definition of "provoked" is left to the treating physician, a DVT in the setting of pelvic surgery or trauma would be considered "provoked"
* Women of child-bearing potential must have a negative pregnancy test prior to treatment on study; breastfeeding should be discontinued if the mother is treated with temsirolimus

  * Women of child-bearing potential and men must agree to use adequate contraception (barrier method of birth control or abstinence; oral contraceptives [also known as "the pill"] are not acceptable) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Patients with a concomitant invasive malignancy or a history of other invasive malignancies, with the exception of non-melanoma skin cancer, are excluded if there is any evidence of other malignancy being present within the past five years; patients are also excluded if their previous cancer treatment contraindicates this protocol therapy
* Patients who have received hormonal therapy or biologic therapy as treatment for endometrial carcinoma
* Patients who have received chemotherapy directed at metastatic or recurrent endometrial carcinoma

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2008-09; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gini Fleming, Principal Investigator — NRG Oncology
Locations (108):
- United States (108):
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Stanford Cancer Institute, Palo Alto, California
  - University of California San Diego, San Diego, California
  - Colorado Gynecologic Oncology Group, Aurora, Colorado
  - University of Colorado Cancer Center - Anschutz Cancer Pavilion, Aurora, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - John B Amos Cancer Center, Columbus, Georgia
  - Memorial University Medical Center, Savannah, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Sudarshan K Sharma MD Limted-Gynecologic Oncology, Hinsdale, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Saint Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Menorah Medical Center, Overland Park, Kansas
  - Radiation Oncology Practice Corporation Southwest, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Shawnee Mission Medical Center-KCCC, Shawnee Mission, Kansas
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - Union Hospital of Cecil County, Elkton, Maryland
  - University of Massachusetts Memorial Health Care, Worcester, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Spectrum Health Big Rapids Hospital, Big Rapids, Michigan
  - Beaumont Hospital-Dearborn, Dearborn, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Green Bay Oncology - Iron Mountain, Iron Mountain, Michigan
  - Allegiance Health, Jackson, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Radiation Oncology Practice Corporation South, Kansas City, Missouri
  - Saint Joseph Health Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Radiation Oncology Practice Corporation - North, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Radiation Oncology Center, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Saint Joseph Oncology Inc, Saint Joseph, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Southwest Gynecologic Oncology Associates Inc, Albuquerque, New Mexico
  - Women's Cancer Care Associates LLC, Albany, New York
  - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - North Shore-LIJ Health System/Center for Advanced Medicine, New Hyde Park, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - University of Cincinnati/Barrett Cancer Center, Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Compass Oncology Rose Quarter, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Black Hills Obstetrics and Gynecology, Rapid City, South Dakota
  - Parkland Memorial Hospital, Dallas, Texas
  - Clements University Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Carilion Clinic Gynecological Oncology, Roanoke, Virginia
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Green Bay Oncology - Oconto Falls, Oconto Falls, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Seventy-three patients were registered to this trial between 9/29/08 and 11/22/10. On 10/19/09 the trial was suspended and the combination arm was permanently closed to accrual because an excess of venous thromboses was noted. The single agent arm continued to the second stage of accrual on 5/24/2010.
Groups:
- Arm 1: Temsirolimus: Temsirolimus IV 25 mg (flat dose) weekly
- Arm 2: Megestrol Acetate+Tamoxifen+ Temsirolimus: Megestrol Acetate (MA) 80 mg bid for three weeks alternating with Tamoxifen (T) 20 mg bid for 3 weeks PLUS Temsirolimus IV 25 mg (flat dose) weekly
Period: Overall Study
Arm/Group | Arm 1: Temsirolimus | Arm 2: Megestrol Acetate+Tamoxifen+ Temsirolimus
Started | 51 | 22
Completed | 50 (Eligible and treated patients) | 21 (Eligible and treated patients)
Not Completed | 1 | 1
Not completed — Ineligible | 0 | 1
Not completed — never treated | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Temsirolimus | Arm 2: Megestrol Acetate+Tamoxifen+ Temsirolimus | Total
Number analyzed (Participants) | 50 | 21 | 71
Age, Customized [Count of Participants; unit: Participants]
  40-49 years | 4 | 0 | 4
  50-59 years | 9 | 6 | 15
  60-69 years | 26 | 10 | 36
  70-79 years | 8 | 3 | 11
  >=80 years | 3 | 2 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 21 | 71
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 1 | 6
  White | 45 | 20 | 65
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Confirmed Objective Tumor Response Using RECIST Version 1.0
Description: RECIST 1.0 defines complete response as the disappearance of all target lesions and non-target lesions and no evidence of new lesions documented by two disease assessments at least 4 weeks apart. Partial response is defined as at least a 30% decrease in the sum of longest dimensions (LD) of all target measurable lesions taking as reference the baseline sum of LD. There can be no unequivocal progression of non-target lesions and no new lesions. Documentation by two disease assessments at least 4 weeks apart is required. In the case where the ONLY target lesion is a solitary pelvic mass measured by physical exam, which is not radiographically measurable, a 50% decrease in the LD is required. These patients will have their response classified according to the definitions stated above. Complete and partial responses are included in the objective tumor response rate.
Time Frame: Radiologic tumor evaluations at baseline and every 6 weeks for the first 24 weeks; then repeated every 12 weeks until disease progression. Repeat after treatment discontinuation if patient was taken off study for reasons other than progression.
Population: Eligible and treated patients
Measure: Number (94% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1: Temsirolimus | Arm 2: Megestrol Acetate+Tamoxifen+ Temsirolimus
Number analyzed (Participants) | 50 | 21
percentage of participants | 22 [11 to 52] | 14.3 [3 to 36]

2. Secondary Outcome: Duration of Overall Survival (OS)
Description: Overall survival is defined as the duration of time from study entry to time of death or the date of last contact.
Time Frame: Every 6 weeks during treatment, then every 3 months for one year.
Population: Eligible and treated patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1: Temsirolimus | Arm 2: Megestrol Acetate+Tamoxifen+ Temsirolimus
Number analyzed (Participants) | 50 | 21
months | 13.3 [9.8 to 20.7] | 9.6 [6.4 to 16.3]

3. Secondary Outcome: Duration of Progression-free Survival (PFS)
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions assessed radiographically and 50% increase if the only target lesion is a solitary pelvic mass measured by physical exam, or unequivocal progression of a non-target lesion, or the appearance of new lesions.
Time Frame: Radiologic tumor evaluations at baseline and every six weeks for the first 24 weeks and then repeated every 12 weeks until disease progression. Repeat after treatment discontinuation if patient was taken off study for reasons other than progression.
Population: Eligible and treated patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1: Temsirolimus | Arm 2: Megestrol Acetate+Tamoxifen+ Temsirolimus
Number analyzed (Participants) | 50 | 21
months | 5.6 [4.0 to 8.2] | 4.2 [1.5 to 6.2]

4. Secondary Outcome: Incidence of Adverse Effects (Grade 3 or Higher) as Assessed by Common Terminology Criteria for Adverse Events Version 3.0
Description: Number of participants with a maximum grade of 3 or higher during the treatment period.
Time Frame: Assessed every 6 weeks while on treatment, 30 days after the last cycle of treatment.
Population: Eligible and treated patients
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Temsirolimus | Arm 2: Megestrol Acetate+Tamoxifen+ Temsirolimus
Number analyzed (Participants) | 50 | 21
Participants | 29 | 15

5. Other Pre Specified Outcome: Number of Participants and Their Levels of Expression of the Candidate Markers
Description: The levels of expression of the candidate markers measured prior to study treatment are tabulated. The expressions being tabulated include immunohistochemical expression of hormone receptors. The hormone receptors are estrogen receptor positive, progesterone receptors-A, progesterone receptor-B, PAKT Positive and PTEN Positive. The associations between the immunohistochemical expression of these biomarkers and between these biomarkers and treatment, outcome or clinical characteristics are reported for future investigation.
Time Frame: Baseline
Population: Eligible and treated patients with primary tumor specimen
Measure: Number; unit: participants
Groups:
- Receptor Analysis: Eligible and treated patients with primary tumor specimen
Arm/Group | Receptor Analysis
Number analyzed (Participants) | 56
participants
  Estrogen Receptor Positive | 20
  Progesterone Receptor Positive | 30
  Progesterone Receptor B Positive | 35
  PAKT Positive | 11
  PTEN Positive | 30

ADVERSE EVENTS:
Time Frame: Assessed every 6 weeks while on treatment, 30 days after the last cycle of treatment, and up to 1 year in follow-up
Arm/Group | Arm 1: Temsirolimus | Arm 2: Megestrol Acetate+Tamoxifen+ Temsirolimus
All-Cause Mortality (participants affected / at risk) | 33/50 | 16/21
Serious Adverse Events (participants affected / at risk) | 18/50 | 13/21
Other Adverse Events (participants affected / at risk) | 50/50 | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Temsirolimus (N=50) | Arm 2: Megestrol Acetate+Tamoxifen+ Temsirolimus (N=21)
Cardiac Arrhythmia - Other (Cardiac disorders) | 1 | 0
Cardiac Ischemia/Infarction (Cardiac disorders) | 0 | 1
Fatigue (General disorders) | 2 | 0
Death No Ctcae Term - Disease Progression Nos (General disorders) | 1 | 2
Death No Ctcae Term - Sudden Death (General disorders) | 0 | 1
Ulceration (Skin and subcutaneous tissue disorders) | 1 | 0
Obstruction, Gi - Small Bowel Nos (Gastrointestinal disorders) | 2 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1
Anorexia (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Joint (Infections and infestations) | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Skin(Cellulitis) (Infections and infestations) | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Urinary Tract Nos (Infections and infestations) | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Abdomen Nos (Infections and infestations) | 1 | 0
Edema: Limb (Blood and lymphatic system disorders) | 0 | 1
Creatinine (Metabolism and nutrition disorders) | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0
Muscle Weakness - Whole Body/Generalized (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain: Extremity-Limb (General disorders) | 0 | 1
Pain: Back (General disorders) | 1 | 0
Dlco (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Obstruction, Gu - Ureter (Renal and urinary disorders) | 1 | 0
Intra-Op Injury: Other (Surgical and medical procedures) | 1 | 0
Thrombosis/Embolism (Vascular Access-Related) (Vascular disorders) | 0 | 1
Thrombosis/Thrombus/Embolism (Vascular disorders) | 2 | 5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Temsirolimus (N=50) | Arm 2: Megestrol Acetate+Tamoxifen+ Temsirolimus (N=21)
Allergic Reaction/Hypersensitivity (Immune system disorders) | 1 | 1
Rhinitis (Immune system disorders) | 2 | 3
Auditory/Ear - Other (Ear and labyrinth disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Neutrophils (Blood and lymphatic system disorders) | 15 | 4
Platelets (Blood and lymphatic system disorders) | 15 | 11
Blood/Bone Marrow - Other (Blood and lymphatic system disorders) | 2 | 0
Leukocytes (Blood and lymphatic system disorders) | 27 | 7
Lymphopenia (Blood and lymphatic system disorders) | 2 | 1
Hemoglobin (Blood and lymphatic system disorders) | 39 | 20
S/N Arrhythmia: Atrial Fibrillation (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Cardiac Arrhythmia - Other (Cardiac disorders) | 1 | 0
S/N Arrhythmia: Sinus Tachycardia (Cardiac disorders) | 0 | 1
Cardiac Ischemia/Infarction (Cardiac disorders) | 0 | 1
Hypertension (Cardiac disorders) | 2 | 0
Lt Ventricular Systolic Dysfunction (Cardiac disorders) | 0 | 1
Hypotension (Cardiac disorders) | 0 | 1
Inr (Vascular disorders) | 0 | 1
Ptt (Vascular disorders) | 1 | 0
Constitutional Symptoms - Other (General disorders) | 0 | 1
Sweating (General disorders) | 1 | 1
Weight Gain (General disorders) | 0 | 2
Fever (General disorders) | 7 | 3
Weight Loss (General disorders) | 8 | 2
Rigors/Chills (General disorders) | 1 | 2
Fatigue (General disorders) | 38 | 18
Insomnia (General disorders) | 4 | 7
Death No Ctcae Term - Disease Progression Nos (General disorders) | 1 | 2
Death No Ctcae Term - Sudden Death (General disorders) | 0 | 1
Nail Changes (Skin and subcutaneous tissue disorders) | 6 | 2
Hair Loss/Alopecia (Scalp Or Body) (Skin and subcutaneous tissue disorders) | 3 | 3
Induration (Skin and subcutaneous tissue disorders) | 0 | 1
Cheilitis (Skin and subcutaneous tissue disorders) | 1 | 1
Wound Complication, Non-Infectious (Skin and subcutaneous tissue disorders) | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 2 | 3
Rash (Skin and subcutaneous tissue disorders) | 27 | 7
Dry Skin (Skin and subcutaneous tissue disorders) | 4 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 10 | 3
Burn (Skin and subcutaneous tissue disorders) | 1 | 0
Flushing (Skin and subcutaneous tissue disorders) | 2 | 1
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 1 | 5
Ulceration (Skin and subcutaneous tissue disorders) | 3 | 2
Hot Flashes (Endocrine disorders) | 2 | 4
Heartburn (Gastrointestinal disorders) | 1 | 2
Mucositis (Functional/Sympt) - Trachea (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 2 | 1
Leak, Gi - Rectum (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Distention (Gastrointestinal disorders) | 3 | 1
Taste Alteration (Gastrointestinal disorders) | 10 | 4
Dry Mouth (Gastrointestinal disorders) | 2 | 2
Mucositis (Functional/Sympt) - Oral Cavity (Gastrointestinal disorders) | 7 | 7
Obstruction, Gi - Small Bowel Nos (Gastrointestinal disorders) | 3 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Mucositis (Clinical Exam) - Oral Cavity (Gastrointestinal disorders) | 10 | 4
Mucositis (Clinical Exam) - Anus (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 13 | 4
Anorexia (Gastrointestinal disorders) | 18 | 4
Dehydration (Gastrointestinal disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 15 | 5
Nausea (Gastrointestinal disorders) | 23 | 3
Diarrhea (Gastrointestinal disorders) | 16 | 8
Hemorrhage, Gu - Vagina (Vascular disorders) | 5 | 0
Hemorrhage, Gi - Varices (Rectal) (Vascular disorders) | 1 | 0
Hemorrhage, Gi - Upper Gi Nos (Vascular disorders) | 0 | 1
Hemorrhage/Pulmonary - Nose (Vascular disorders) | 3 | 5
Hemorrhage, Gu - Ureter (Vascular disorders) | 1 | 0
Petechiae (Vascular disorders) | 0 | 1
Hemorrhage/Bleeding - Other (Vascular disorders) | 2 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Upper Airway Nos (Infections and infestations) | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Paranasal (Infections and infestations) | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Lung(Pneumonia) (Infections and infestations) | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Eye Nos (Infections and infestations) | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Soft Tissue Nos (Infections and infestations) | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Joint (Infections and infestations) | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Blood (Infections and infestations) | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Small Bowel Nos (Infections and infestations) | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Oral Cavity-Gums (Infections and infestations) | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Skin(Cellulitis) (Infections and infestations) | 1 | 1
Inf Unknown Anc: Lung (Pneumonia) (Infections and infestations) | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Urinary Tract Nos (Infections and infestations) | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Abdomen Nos (Infections and infestations) | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Ungual (Nails) (Infections and infestations) | 1 | 0
Infection - Other (Infections and infestations) | 2 | 0
Colitis, Infectious (Eg.C. Difficile) (Infections and infestations) | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Nerve-Peripheral (Infections and infestations) | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Bronchus (Infections and infestations) | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Mucosa (Infections and infestations) | 0 | 1
Inf Unknown Anc: Upper Airway Nos (Infections and infestations) | 1 | 0
Inf W/Nml Or Gr 1 Or 2 Anc: Sinus (Infections and infestations) | 0 | 1
Inf Unknown Anc: Urinary Tract Nos (Infections and infestations) | 0 | 1
Inf Unknown Anc: Skin (Cellulitis) (Infections and infestations) | 0 | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Kidney (Infections and infestations) | 1 | 0
Lymphedema-Related Fibrosis (Blood and lymphatic system disorders) | 0 | 1
Edema: Trunk/Genital (Blood and lymphatic system disorders) | 0 | 1
Edema: Limb (Blood and lymphatic system disorders) | 16 | 10
Edema: Head And Neck (Blood and lymphatic system disorders) | 2 | 3
Ast (Metabolism and nutrition disorders) | 5 | 1
Gfr (Metabolism and nutrition disorders) | 0 | 1
Metabolic/Laboratory - Other (Metabolism and nutrition disorders) | 1 | 2
Cholesterol,serum High (Metabolism and nutrition disorders) | 19 | 7
Creatinine (Metabolism and nutrition disorders) | 9 | 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 7 | 6
Alt (Metabolism and nutrition disorders) | 4 | 1
Alkaline Phosphatase (Metabolism and nutrition disorders) | 7 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 6 | 4
Hypertriglyceridemia (Metabolism and nutrition disorders) | 20 | 7
Bicarbonate, Serum-Low (Metabolism and nutrition disorders) | 1 | 0
Hypernatremia (Metabolism and nutrition disorders) | 2 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 8 | 3
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 9 | 3
Hypokalemia (Metabolism and nutrition disorders) | 10 | 4
Hypoglycemia (Metabolism and nutrition disorders) | 2 | 2
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 3 | 3
Musculoskeletal/St: Other (Musculoskeletal and connective tissue disorders) | 1 | 1
Fracture (Musculoskeletal and connective tissue disorders) | 1 | 1
Extremity-Upper (Function) (Musculoskeletal and connective tissue disorders) | 2 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle Weakness - Whole Body/Generalized (Musculoskeletal and connective tissue disorders) | 3 | 2
Syncope (Nervous system disorders) | 1 | 0
Psychosis (Nervous system disorders) | 0 | 1
Mood Alteration - Depression (Nervous system disorders) | 2 | 1
Mood Alteration - Anxiety (Nervous system disorders) | 4 | 1
Mood Alteration - Agitation (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 2
Speech Impairment (Nervous system disorders) | 1 | 0
Irritability (Nervous system disorders) | 0 | 1
Confusion (Nervous system disorders) | 2 | 0
Memory Impairment (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 3 | 4
Neuropathy-Sensory (Nervous system disorders) | 7 | 1
Ocular/Visual - Other (Eye disorders) | 1 | 0
Watery Eye (Eye disorders) | 1 | 0
Dry Eye (Eye disorders) | 1 | 0
Pain - Other (General disorders) | 2 | 4
Pain: Urethra (General disorders) | 0 | 1
Pain: Breast (General disorders) | 0 | 1
Pain: Chest /Thorax Nos (General disorders) | 1 | 1
Pain: Chest Wall (General disorders) | 1 | 1
Pain: Throat/Pharynx/Larynx (General disorders) | 2 | 1
Pain: Head/Headache (General disorders) | 8 | 4
Pain: Neck (General disorders) | 0 | 1
Pain: Extremity-Limb (General disorders) | 6 | 3
Pain: Buttock (General disorders) | 1 | 0
Pain: Back (General disorders) | 9 | 2
Pain: Joint (General disorders) | 4 | 3
Pain: Kidney (General disorders) | 1 | 0
Pain: Bladder (General disorders) | 1 | 0
Pain: Pain Nos (General disorders) | 1 | 2
Pain: Stomach (General disorders) | 1 | 1
Pain: Oral Cavity (General disorders) | 2 | 0
Pain: Dental/Teeth/Peridontal (General disorders) | 0 | 1
Pain: Abdominal Pain Nos (General disorders) | 12 | 6
Pain: Muscle (General disorders) | 4 | 2
Pulmonary: Other (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Nasal/Paranasal Reactions (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Voice Changes (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Fev1 (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 5
Dlco (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 14 | 13
Renal/Genitourinary - Other (Renal and urinary disorders) | 1 | 0
Stricture, Anastomotic, Gu - Ureter (Renal and urinary disorders) | 0 | 1
Cystitis (Renal and urinary disorders) | 1 | 0
Obstruction, Gu - Ureter (Renal and urinary disorders) | 1 | 0
Incontinence, Urinary (Renal and urinary disorders) | 1 | 1
Renal Failure (Renal and urinary disorders) | 0 | 1
Urinary Frequency (Renal and urinary disorders) | 1 | 2
Breast (Reproductive system and breast disorders) | 1 | 0
Vaginal Dryness (Reproductive system and breast disorders) | 1 | 0
Sexual/Reproductive Function: Other (Reproductive system and breast disorders) | 1 | 0
Flu-Like Syndrome (General disorders) | 0 | 1
Artery Injury - Extremity-Lower (Vascular disorders) | 0 | 1
Thrombosis/Embolism (Vascular Access-Related) (Vascular disorders) | 0 | 1
Thrombosis/Thrombus/Embolism (Vascular disorders) | 3 | 5
Phlebitis (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
The combination arm was closed after the first stage of accrual due to an excess of venous thromboses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-12-22): https://cdn.clinicaltrials.gov/large-docs/86/NCT00729586/Prot_SAP_000.pdf